CLINICAL TRIAL: NCT00817479
Title: Tumor Gene Expression Before and After Intraoperative Dexamethasone in Women With Ovarian Cancer
Brief Title: Tumor Gene Expression in Women With Ovarian Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 11892A
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Results first posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-06

CONDITIONS: Ovarian Cancer
Keywords: Subject has intraabdominal disease either proven or strongly; suspected to be ovarian or primary peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator): 20 mg of dexamethasone
  Interventions: Drug: Dexamethasone
- Placebo [Saline] (Placebo Comparator): Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — 20 MG OF DEXAMETHASONE OR PLACEBO
  Arms: Dexamethasone
Drug: Placebo — Placebo saline
  Other Names: Saline Placebo
  Arms: Placebo [Saline]

SUMMARY:
The study objective is to compare changes in expression of glucocorticoid-induced genes that may be involved in cell survival signaling in the tumors of ovarian cancer patients before and after an intraoperative dose of 20mg dexamethasone.

DETAILED DESCRIPTION:
This trial will examine the upregulation of dexamethasone-inducible genes in the tumors of ovarian cancer patients undergoing surgical debulking. A core biopsy of tumor will be taken at the first opportune time during surgery. Dexamethasone 20 mg IV will then be administered, and a second biopsy taken 30 minutes later. Samples at two and four hours later will also be obtained if surgery is still in progress and biopsiable tumor remains. Tissue will be snap-frozen. Subsequently tumor will be microdissected out from stroma, and tumor RNA will be extracted for gene expression profiling. Sixteen patients with epithelial ovarian cancer receiving dexamethasone will be studied, and an additional eight patients with epithelial ovarian cancer will receive a small saline (placebo) injection and serve as controls. Enrollment is limited to those patients with a serum albumin of at least 3.0 g/dL to minimize any theoretical adverse effect of a single dose of dexamethasone on wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Subject has intraabdominal disease either proven or strongly suspected to be ovarian or primary peritoneal cancer, and will be undergoing surgical debulking.
* Subject is not allergic to dexamethasone, and there is no obvious medical contraindication to dexamethasone.
* Subjects with diabetes requiring drug therapy are excluded.
* Subject is not currently receiving glucocorticoid therapy
* Nasal steroids (e.g. Flonase) are permitted
* Subject understands that this protocol does not have therapeutic intent
* Preoperative serum albumin at least 3.0 mg/dL
* Negative serum or urine pregnancy test in women of childbearing potential
* Signed informed consent

Exclusion Criteria:

* Males do not get ovarian cancer and therefore will not be included in this trial.
* Patients of all ethnic backgrounds are eligible and will be encouraged to enroll. However we do not expect differences based on ethnicity, and this small study will not therefore be powered to make conclusions about ethnic differences in induction of GR-regulated genes with dexamethasone.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gini Fleming, MD, Study Chair — Gralla, R. J., Osoba, D., Kris, M. G., Kirkbride, P., Hesketh, P. J., et al.: Recommendations for the use of antiemetics: evidence-based, clinical practice guidelines. American Society of Clinical Oncology. J Clin Oncol 1999; 17(9): 2971-94.
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Melhem A, Yamada SD, Fleming GF, Delgado B, Brickley DR, Wu W, Kocherginsky M, Conzen SD. Administration of glucocorticoids to ovarian cancer patients is associated with expression of the anti-apoptotic genes SGK1 and MKP1/DUSP1 in ovarian tissues. Clin Cancer Res. 2009 May 1;15(9):3196-204. doi: 10.1158/1078-0432.CCR-08-2131. Epub 2009 Apr 21. PMID 19383827

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between July 2003 and September 2007 through the Gynecologic Oncology Clinic at the University of Chicago subject to the inclusion and exclusion criteria described in the registration record.
Groups:
- Placebo: Placebo [saline]
- Dexamethasone: 20 mg dexamethasone IV push
Period: Overall Study
Arm/Group | Placebo | Dexamethasone
Started | 6 | 14
Completed | 5 | 13
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dexamethasone | Total
Number analyzed (Participants) | 6 | 14 | 20
Age, Continuous [Median (Full Range); unit: years] | 61 [46 to 80] | 53.5 [44 to 73] | 56 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 20
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Increase in SGK1 mRNA Expression Level
Description: Increase in SGK1 mRNA expression level is calculated as fold change = post / pre
Time Frame: >= 30 min
Population: Eighteen of the 20 randomized patients received treatment. Eight of the treated patients were unevaluable because there was not enough tissue available during surgery for experimental studies; the remaining 10 patients had adequate tissue samples at baseline and at least at 30 minutes following dexamethasone/normal saline administration.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Placebo | Dexamethasone
Number analyzed (Participants) | 5 | 5
fold change | 1.5 (0.4) | 6.1 (2.6)

2. Primary Outcome: Increase in MKP1/DuSP1 mRNA Expression Level
Description: Increase in MKP1/DuSP1 mRNA expression level is calculated as fold change = post / pre
Time Frame: >= 30 min
Population: as for outcome 1
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Placebo | Dexamethasone
Number analyzed (Participants) | 5 | 5
fold change | 1.1 (0.4) | 8.2 (2.9)

ADVERSE EVENTS:
Time Frame: Intra-operative assessment. Patients were not followed after surgery.
Arm/Group | Placebo | Dexamethasone
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/14
Other Adverse Events (participants affected / at risk) | 0/6 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes